CLINICAL TRIAL: NCT01657266
Title: Phase 2 Randomized, Double-blind Clinical Trial to Evaluate Efficacy and Safety of the Ophthalmic Solution PRO-155 Versus Nevanac 0.1% Ophthalmic Solution in Post Phacoemulsification Patients
Brief Title: Efficacy and Safety of PRO-155 Versus Nevanac in Post Phacoemulsification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH155-0412/II
Record Dates: First submitted 2012-07-19; First posted 2012-08-06 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-02

CONDITIONS: Cataract; Phacoemulsification Cataract Surgery
Keywords: bromfenac; nepafenac; cataract; phacoemulsification cataract surgery
MeSH Terms: conditions — Cataract | interventions — nepafenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRO-155 (Experimental): Bromfenac 0.09% (0.9mg/mL) Ophthalmic solution Pre-medication: 1 drop each 15 minutes during 1 hour before surgery in the affected eye
  Maintenance therapy: 1 drop 3 times a day for 30 days
  Interventions: Drug: PRO-155
- Nevanac (Active Comparator): Nepafenac 0.1% (1mg/mL) Ophthalmic Suspension
  Pre-medication: 1 drop each 15 minutes during 1 hour before surgery in the affected eye
  Maintenance therapy: 1 drop 3 times a day for 30 days
  Interventions: Drug: Nevanac

INTERVENTIONS:
Drug: PRO-155 — Pre-medication (before surgery) and maintenance treatment.
  Arms: PRO-155
Drug: Nevanac — Pre-medication (before surgery) and maintenance treatment.
  Arms: Nevanac

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of the ophthalmic solution PRO-155 in patients post phacoemulsification.

DETAILED DESCRIPTION:
Postsurgical inflammation is an inevitable condition after cataract surgery. The use of non-steroidal anti-inflammatory drugs is a safe option for treating ocular inflammation.

This is a phase II randomized double-blind clinical trial. The aim is to compare and to evaluate efficacy and safety of two ophthalmic solutions in patients post phacoemulsification. Patients will be randomized to receive either PRO-155 or Nevanac for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years who require cataract surgery
* Both genders
* Provide informed consent
* Normal Laboratory results

Exclusion Criteria:

* Patients with visual acuity of 20/40 or less in the contralateral eye of the surgery
* Patients with any trans-surgical complication
* Patients with a cataract >NC4, C4 or P4 classified with the system LOCS
* Patients with any active corneal pathology
* Patients under any steroidal treatment (topic, systemic or inhaled)14 days prior surgery or NSAIDs 7 days before the surgery (except low-dose aspirin)
* Patients with IOP <5 or >21 mmHg
* Patients that have ocular pain, cellularity or flare at the moment of selection
* Patients with ocular exfoliation, trauma or any inflammatory disease
* Patients with diabetic retinopathy that need treatment or uncontrolled diabetes mellitus
* Patients who are planning cataract surgery of the contralateral eye 14 days after surgery of the study eye
* Patients with history of hypersensitivity or contraindication for any drug used in the study
* Patients under anticoagulant treatment
* Contact lens users
* Pregnant patients, at risk of pregnancy or breastfeeding
* Patients without birth control treatment
* Patients with any active toxicomania (alcoholism, cigarette, cannabis or others)
* Patients who had participated in any clinical trial in the last 90 days
* Legal or mentally disabled patients who could not give informed consent
* Patients who cannot comply with all study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo M. Baiza-Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The personal data were collected and analyzed according to confidentiality policy.

REFERENCES:
- See also: Palacio C, et al. Bromfenac 0.09% bioavailability in aqueous humor, prophylactic effect on cystoid macular edema, and clinical signs of ocular inflammation after phacoemulsification in a Mexican population. Clinical Ophthalmology 2016;10:233-237 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4734805/pdf/opth-10-233.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 160 subjects were recruited, 12 of whom were excluded, 10 because they did not meet the selection criteria and 2 refused to participate. The remaining 148 were randomly assigned to one of the 2 study groups, 73 to bromfenac and 75 to napaphenac.
Groups:
- PRO-155: Bromfenac 0.09% (0.9mg/mL) Ophthalmic solution
  Pre-medication: 1 drop each 15 minutes during 1 hour before surgery in the affected eye
  Maintenance therapy: 1 drop 3 times a day for 30 days
  PRO-155: Pre-medication (before surgery) and maintenance treatment.
- Nevanac: Nepafenac 0.1% (1mg/mL) Ophthalmic Suspension
  Pre-medication: 1 drop each 15 minutes during 1 hour before surgery in the affected eye
  Maintenance therapy: 1 drop 3 times a day for 30 days
  Nevanac: Pre-medication (before surgery) and maintenance treatment.
Period: Overall Study
Arm/Group | PRO-155 | Nevanac
Started | 73 | 75
Completed | 69 | 70
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 2 | 3

BASELINE CHARACTERISTICS:
Population: Mexican patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-155 | Nevanac | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (11.1) | 68.0 (9.5) | 67.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 28 | 31 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 70 | 139
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 69 | 70 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cellularity in Anterior Chamber
Description: Change from Percentage of Cellularity in anterior chamber after 30 days of treatment.
Time Frame: day 30
Population: Mexican patients patients who underwent cataract surgery in only 1 eye, by phacoemulsification with intraocular lens implantation.
Measure: Number; unit: Percentage of Cellularity
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
Percentage of Cellularity
  Day 1 | 64.2 | 64.3
  Day 30 | 0 | 0
Statistical Analysis 1: Comparison: PRO-155; Test type: Superiority or Other; p = 1.00, Pearson´s Chi-square test

2. Primary Outcome: Flare in Anterior Chamber
Description: Percentage of Participants with flare in anterior chamber after 30 days of treatment
Time Frame: day 30
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants with flare
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
Percentage of Participants with flare
  Day 1 | 31.4 | 31.5
  Day 30 | 0 | 0

3. Secondary Outcome: Percentage of Patients Without Ocular Pain
Description: percentage of patients without pain, would be measured using the Visual Analog Pain Scale
Time Frame: day 30
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
percentage of patients
  Day 1 | 6.1 | 5.7
  Day 30 | 1.5 | 1.6

4. Secondary Outcome: Mean Aqueous Concentration of Intervention Drug
Description: a nurse was instructed to instill five drops of the research product into each patient's eye in the hour before surgery. The concentration of the drug was determined for aqueous humor sample (0.15 mL) with a 30-gauge needle on a TB syringe after completion of the paracentesis. The paracentesis was performed after first incision during the phacoemulsification.
Time Frame: before surgery
Population: We enrolled patients of both sexes (aged >18 years) with a diagnosis of cataract according to the Lens Opacities Classification System III ≤ NC4, C4 and, P4 in one eye were eligible for enrollment. Eligible patients must have had a best-corrected visual acuity of 6/60 (20/200) Snellen score.
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
Number analyzed (eyes) | 69 | 70
ng/mL | 207.5 (152.3) | 314.4 (146.5)

5. Other Pre Specified Outcome: Epithelial Defects Detected With Fluorescein
Description: The percentage of patients presenting epithelial defects with fluorescein staining will be evaluated
Time Frame: measurements will be made at days 1, 5, 7 and 30
Population: as for outcome 1
Measure: Number; unit: percentage of patients with defects
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
percentage of patients with defects
  Day 1 | 54.4 | 78.5
  Day 7 | 32.5 | 64.4
  Day 15 | 15.6 | 36.1
  Day 30 | 6 | 8.5

6. Other Pre Specified Outcome: Epithelial Defects Detected With Green Lissamine
Description: the percentage of patients presenting epithelial defects evaluated with green lysine will be reported
Time Frame: measurements will be made at days 1, 5, 7 and 30
Population: Mexican patients who underwent cataract surgery in only 1 eye, by phacoemulsification with intraocular lens implantation.
Measure: Number; unit: percentage of patients with defects
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
percentage of patients with defects
  Day 1 | 62.5 | 86
  Day 7 | 41.4 | 67.3
  Day 15 | 21.6 | 57.4
  Day 30 | 14.8 | 28.2

7. Other Pre Specified Outcome: Intraocular Pressure
Description: Change from Baseline in the intraocular pressure after 30 days of treatment
Time Frame: day 30
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
mmHg
  Day 0 | 14.07 (1.82) | 14.23 (1.90)
  Day 1 | 14.66 (2.61) | 15.83 (2.77)
  Day 7 | 14.13 (1.97) | 14.54 (1.85)
  Day 15 | 13.81 (1.64) | 13.91 (2.03)
  Day 30 | 14.10 (1.78) | 13.77 (1.97)

8. Other Pre Specified Outcome: Retinal Thickness
Description: Change from Baseline in retinal thickness after 30 days of treatment. A third measurement will be done at 60 day after day surgery.
Time Frame: day 30 and 60
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | PRO-155 | Nevanac
Number analyzed (Participants) | 69 | 70
μm
  field A1 day 0 | 247.24 (32.90) | 250.87 (34.42)
  field A1 day 30 | 252.06 (24.95) | 264.08 (34.10)
  field A1 day 60 | 254.06 (2.78) | 260.13 (33.93)

ADVERSE EVENTS:
Time Frame: Interval of 30 days of intervention in which adverse events could occur, included in the treatment period (January 2014-2015)
Description: During the pharmacological intervention period, in each visit, the principal investigator asked information about adverse events:
  1. Serious or No serious
  2. Severity: mild, moderate, severe
  3. relation with study drug or not
Arm/Group | PRO-155 | Nevanac
Serious Adverse Events (participants affected / at risk) | 0/73 | 2/75
Other Adverse Events (participants affected / at risk) | 5/73 | 2/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-155 (N=73) | Nevanac (N=75)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1) — This serious adverse event occurred during the systematic assessment. The event was not related with the pharmacological intervention.
central retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) — This serious adverse event occurred during systematic assessment. The adverse event was not related with the pharmacological intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-155 (N=73) | Nevanac (N=75)
fall from their own height (Vascular disorders) | 0 (0) | 1 (1) — The mild adverse event does not have relationship with the study drug.
Cystoid macular edema (Eye disorders) | 1 (1) | 0 (0) — This moderate adverse event does not relationship with the study drug. The clinically significant cystoid macular edema occurs after cataract surgery.
Traumatic corneal desepithelization (Eye disorders) | 1 (1) | 0 (0) — This moderate event does not have relationship with the study drug. The patient presented an accidental ocular injure.
Posterior Capsular Rupture (Eye disorders) | 1 (1) | 0 (0) — This mild adverse event does not relationship with the study drug. The posterior capsular rupture occurs after cataract surgery.
viral conjunctivitis (Eye disorders) | 1 (1) | 0 (0) — This severe adverse event does not have relationship with the study drug. This patient had hypothyroidism like concomitant disease, this clinical condition would be able to increase the risk to have an infectious disease.
Inflammatory cells in the corneal endothelium (Eye disorders) | 1 (1) | 0 (0) — This moderate adverse event does not have relationship with the study drug. The presence of inflammatory cells in the corneal endothelium is related to cataract surgery procedure.
intraocular lens exchange (Eye disorders) | 0 (0) | 1 (1) — This adverse event does not have relationship with the study drug. The reason of intraocular lens exchange was: error in the intraocular lens power calculation.

LIMITATIONS AND CAVEATS:
The study was performed according to the clinical protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information is confidential and exclusive property of the sponsor. Information can be revealed only to my staff and regulatory agencies or ethics committee.

All the information from this protocol is confidential and exclusive property of the sponsor, it can not be revealed without written consent from the sponsor.